CLINICAL TRIAL: NCT05589467
Title: What Are the Effects of Potatoes, Utilizing Specific Cooking Methods, on Blood Pressure in Hypertensive Persons With and Without Type II Diabetes Who Follow the DASH Diet for 6 Weeks?
Brief Title: Effects of Potatoes on Blood Pressure in Persons With and Without Type 2 Diabetes Who Follow the DASH Diet for 6 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, Shannon Galyean, Assistant Professor/Registered Dietitian Nutritionist, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB2019-880
Record Dates: First submitted 2022-09-16; First posted 2022-10-21 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes; Blood Pressure
Keywords: DASH diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DASH Diet and Fried Potatoes (Experimental): DASH-FP (fried potatoes) group
  Interventions: Other: DASH-FP
- DASH Diet and Non-Fried Potatoes (Experimental): DASH-NFP (non-fried potatoes) group
  Interventions: Other: DASH-NFP
- DASh Diet and No Potatoes (Experimental): DASH-NP (no potatoes) group
  Interventions: Other: Control

INTERVENTIONS:
Other: DASH-FP — Dash diet with only fried potatoes
  Arms: DASH Diet and Fried Potatoes
Other: DASH-NFP — Dash diet with only non-fried potatoes
  Arms: DASH Diet and Non-Fried Potatoes
Other: Control — Dash diet with no potatoes
  Arms: DASh Diet and No Potatoes

SUMMARY:
This study will be a randomized controlled intervention study that will collect pre-intervention and post-intervention anthropometric health data of men and women aged 18-65 years who have type 2 diabetes and who do not have type 2 diabetes. The information collected will be analyzed and used to compare to the post intervention. 12 participants who have type 2 diabetes and 12 participants who do not have type 2 diabetes will be randomized into either the DASH-FP (fried potatoes), DASH-NFP (non-fried potatoes) or DASH-NP (no potatoes) groups, stratifying by sex (male or female) and age range (18 to less than 35, 35 to less than 66 years old) in blocks of three.

DETAILED DESCRIPTION:
Subjects will follow the DASH diet for 2 weeks to establish baseline blood pressure and then will be randomized to a 4-week intervention study with assigned dietary patterns (DASH-NP as a control diet, DASH-FP diet with only fried potatoes, or DASH-NFP diet with only non-fried potatoes) in accordance with the protocol given above. Before intervention, each group will receive a cooking demonstrations, samples, and recipes to show the correct preparation method and seasoning ingredient to use according to each treatment group. The control group will receive a cooking demonstration including DASH diet recipes without potatoes. Potatoes will be provided for participants in the potato groups allowing for one serving a day of potatoes prepared according to their treatment group.

The control diet will be the standard DASH diet but with no potatoes. DASH-FP will include 5 servings of fried potatoes each week. DASH-NFP will include 5 servings of non-fried potatoes each week. Participants will be instructed to maintain the broad requirements of the DASH diet on their own. A 7-day menu cycle from the DASH-Sodium study for each dietary pattern at different energy levels will be used as the basis for the recommended diets. There will be weekly contact with the participants in which the DASH diet will be reinforced. The goal of the weekly sessions will be to assist participants in learning how to buy and prepare the appropriate foods according to their dietary pattern, to enhance their motivation to choose to eat those foods, and to overcome obstacles to following the diet.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

-Well controlled type 2 diabetes as diagnosed by a physician, which is managed by diet and exercise alone or any diabetes medication(s) other than insulin; clinically stable.

Group 2:

-No diagnosis of type 2 diabetes

Group 1 and 2 Exclusion Criteria:

* Use of tobacco
* Self-reported history of chronic diseases other than type 2 diabetes (e.g., cardiovascular, etc.)
* Evidence of severe diabetic complications (such as proliferative retinopathy or diabetic nephropathy)
* Uncontrolled hypertension
* Use of oral steroids, hormone replacement therapy
* Individuals with blood pressure ≥160/100, or HbA1c ≥9%
* Individuals with allergy to potatoes
* Pregnant or lactating
* Individuals on insulin therapy
* Any alcohol or drug dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Systolic and Diastolic blood pressure in mmHg | at baseline
  After the subject has rested for five minutes in a sitting position, blood pressure measurements will be taken, using an Omron IntelliSense® Blood Pressure Monitor using an arm cuff suitable for the body size. Three readings will be taken at five-minute intervals and the average of the three measurements used.
Systolic and Diastolic blood pressure in mmHg | 2 weeks
  After the subject has rested for five minutes in a sitting position, blood pressure measurements will be taken, using an Omron IntelliSense® Blood Pressure Monitor using an arm cuff suitable for the body size. Three readings will be taken at five-minute intervals and the average of the three measurements used.
Systolic and Diastolic blood pressure in mmHg | 6 weeks
  After the subject has rested for five minutes in a sitting position, blood pressure measurements will be taken, using an Omron IntelliSense® Blood Pressure Monitor using an arm cuff suitable for the body size. Three readings will be taken at five-minute intervals and the average of the three measurements used.
Body mass index in kg/m^2 | at baseline
  weight in kg and height in meters will be used to calculate BMI
Waist circumference in inches | at baseline
  A certified non-stretch tape measure will be used to measure waist circumference (WC) at the natural waist (mid-way between the 10th rib and the ileac crest) as recommended by the World Health Organization and hip circumference over the widest point over the buttocks to the nearest centimeter.
Waist circumference in inches | 2 weeks
  A certified non-stretch tape measure will be used to measure waist circumference (WC) at the natural waist (mid-way between the 10th rib and the ileac crest) as recommended by the World Health Organization and hip circumference over the widest point over the buttocks to the nearest centimeter.
Waist circumference in inches | 6 weeks
  A certified non-stretch tape measure will be used to measure waist circumference (WC) at the natural waist (mid-way between the 10th rib and the ileac crest) as recommended by the World Health Organization and hip circumference over the widest point over the buttocks to the nearest centimeter.
body composition in body fat percentage | at baseline
  Body composition (fat and lean body mass) will be measured by bioelectric impedance using a Tanita scale (model SC-331S Tanita, Tokyo, Japan).
body composition in body fat percentage | 2 weeks
  Body composition (fat and lean body mass) will be measured by bioelectric impedance using a Tanita scale (model SC-331S Tanita, Tokyo, Japan).
body composition in body fat percentage | 6 weeks
  Body composition (fat and lean body mass) will be measured by bioelectric impedance using a Tanita scale (model SC-331S Tanita, Tokyo, Japan).
weight in lbs | at baseline
  Weight will be measure to the nearest 0.1lb
weight in lbs | 2 weeks
  Weight will be measure to the nearest 0.1 lb
weight in lbs | 6 weeks
  Weight will be measure to the nearest 0.1 lb
height in centimeters | at baseline
  Height will be measured to the nearest 0.1 cm using a stadiometer.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Galyean, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International Diabetes Federation. IDF Diabetes Atlas, 9th Edn. Brussels, Belgium: International Diabetes Federation, 2019. http://www.diabetesatlas.org
- [Background] Gurushankar Govindarajan, James R Sowers, Craig S Stump (2016) Volume 2, Issue 1 Hypertension and Diabetes Mellitus https://doi.org/10.15420/ecr.2006.1.21
- [Background] Aljuraiban GS, Pertiwi K, Stamler J, Chan Q, Geleijnse JM, Van Horn L, Daviglus ML, Elliott P, Oude Griep LM; INTERMAP Research Group. Potato consumption, by preparation method and meal quality, with blood pressure and body mass index: The INTERMAP study. Clin Nutr. 2020 Oct;39(10):3042-3048. doi: 10.1016/j.clnu.2020.01.007. Epub 2020 Jan 22. PMID 32037285
- [Background] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Background] Azadbakht L, Fard NR, Karimi M, Baghaei MH, Surkan PJ, Rahimi M, Esmaillzadeh A, Willett WC. Effects of the Dietary Approaches to Stop Hypertension (DASH) eating plan on cardiovascular risks among type 2 diabetic patients: a randomized crossover clinical trial. Diabetes Care. 2011 Jan;34(1):55-7. doi: 10.2337/dc10-0676. Epub 2010 Sep 15. PMID 20843978
- [Background] Azadbakht L, Mirmiran P, Esmaillzadeh A, Azizi T, Azizi F. Beneficial effects of a Dietary Approaches to Stop Hypertension eating plan on features of the metabolic syndrome. Diabetes Care. 2005 Dec;28(12):2823-31. doi: 10.2337/diacare.28.12.2823. PMID 16306540
- [Background] Beals, K. A. (2019). Potatoes, Nutrition and Health. American Journal of Potato Research, 96(2), 102-110. doi:10.1007/s12230-018-09705-4
- [Background] Berraho M, El Achhab Y, Benslimane A, El Rhazi K, Chikri M, Nejjari C. Hypertension and type 2 diabetes: a cross-sectional study in Morocco (EPIDIAM Study). Pan Afr Med J. 2012;11:52. Epub 2012 Mar 20. PMID 22593788
- [Background] Challa, H. J., Ameer, M. A., & Uppaluri, K. R. (2020). DASH Diet (Dietary Approaches to Stop Hypertension). In StatPearls. Treasure Island (FL): StatPearls Publishing Copyright © 2020, StatPearls Publishing LLC. 35 45 44
- [Background] Challa, H. J., Tadi, P., & Uppaluri, K. R. (2019). DASH Diet (Dietary Approaches to Stop Hypertension): StatPearls Publishing, Treasure Island (FL).
- [Background] Chen G, McAlister FA, Walker RL, Hemmelgarn BR, Campbell NR. Cardiovascular outcomes in framingham participants with diabetes: the importance of blood pressure. Hypertension. 2011 May;57(5):891-7. doi: 10.1161/HYPERTENSIONAHA.110.162446. Epub 2011 Mar 14. PMID 21403089
- [Background] Cheung BM, Li C. Diabetes and hypertension: is there a common metabolic pathway? Curr Atheroscler Rep. 2012 Apr;14(2):160-6. doi: 10.1007/s11883-012-0227-2. PMID 22281657
- [Background] Cook NR, Cutler JA, Obarzanek E, Buring JE, Rexrode KM, Kumanyika SK, Appel LJ, Whelton PK. Long term effects of dietary sodium reduction on cardiovascular disease outcomes: observational follow-up of the trials of hypertension prevention (TOHP). BMJ. 2007 Apr 28;334(7599):885-8. doi: 10.1136/bmj.39147.604896.55. Epub 2007 Apr 20. PMID 17449506
- [Background] de Paula TP, Steemburgo T, de Almeida JC, Dall'Alba V, Gross JL, de Azevedo MJ. The role of Dietary Approaches to Stop Hypertension (DASH) diet food groups in blood pressure in type 2 diabetes. Br J Nutr. 2012 Jul 14;108(1):155-62. doi: 10.1017/S0007114511005381. Epub 2011 Dec 6. PMID 22142820
- [Background] Drewnowski A. The Nutrient Rich Foods Index helps to identify healthy, affordable foods. Am J Clin Nutr. 2010 Apr;91(4):1095S-1101S. doi: 10.3945/ajcn.2010.28450D. Epub 2010 Feb 24. PMID 20181811
- [Background] Ferrannini E, Cushman WC. Diabetes and hypertension: the bad companions. Lancet. 2012 Aug 11;380(9841):601-10. doi: 10.1016/S0140-6736(12)60987-8. PMID 22883509
- [Background] Obarzanek E, Sacks FM, Vollmer WM, Bray GA, Miller ER 3rd, Lin PH, Karanja NM, Most-Windhauser MM, Moore TJ, Swain JF, Bales CW, Proschan MA; DASH Research Group. Effects on blood lipids of a blood pressure-lowering diet: the Dietary Approaches to Stop Hypertension (DASH) Trial. Am J Clin Nutr. 2001 Jul;74(1):80-9. doi: 10.1093/ajcn/74.1.80. PMID 11451721
- [Background] Halton TL, Willett WC, Liu S, Manson JE, Stampfer MJ, Hu FB. Potato and french fry consumption and risk of type 2 diabetes in women. Am J Clin Nutr. 2006 Feb;83(2):284-90. doi: 10.1093/ajcn/83.2.284. PMID 16469985
- [Background] Hashemi R, Rahimlou M, Baghdadian S, Manafi M. Investigating the effect of DASH diet on blood pressure of patients with type 2 diabetes and prehypertension: Randomized clinical trial. Diabetes Metab Syndr. 2019 Jan-Feb;13(1):1-4. doi: 10.1016/j.dsx.2018.06.014. Epub 2018 Jun 21. PMID 30641678
- [Background] He FJ, MacGregor GA. Effect of modest salt reduction on blood pressure: a meta-analysis of randomized trials. Implications for public health. J Hum Hypertens. 2002 Nov;16(11):761-70. doi: 10.1038/sj.jhh.1001459. PMID 12444537
- [Background] Heller, M. (2011). The DASH Diet Action Plan: Proven to Lower Blood Pressure and Cholesterol Without Medication: Grand Central Publishing.
- [Background] Houston MC, Harper KJ. Potassium, magnesium, and calcium: their role in both the cause and treatment of hypertension. J Clin Hypertens (Greenwich). 2008 Jul;10(7 Suppl 2):3-11. doi: 10.1111/j.1751-7176.2008.08575.x. PMID 18607145
- [Background] Hu G, Jousilahti P, Tuomilehto J. Joint effects of history of hypertension at baseline and type 2 diabetes at baseline and during follow-up on the risk of coronary heart disease. Eur Heart J. 2007 Dec;28(24):3059-66. doi: 10.1093/eurheartj/ehm501. Epub 2007 Nov 2. PMID 17981826
- [Background] Huang M, Zhuang P, Jiao J, Wang J, Chen X, Zhang Y. Potato consumption is prospectively associated with risk of hypertension: An 11.3-year longitudinal cohort study. Clin Nutr. 2019 Aug;38(4):1936-1944. doi: 10.1016/j.clnu.2018.06.973. Epub 2018 Jul 2. PMID 30025746
- [Background] Johnston EA, Petersen KS, Kris-Etherton PM. Daily intake of non-fried potato does not affect markers of glycaemia and is associated with better diet quality compared with refined grains: a randomised, crossover study in healthy adults. Br J Nutr. 2020 May 14;123(9):1032-1042. doi: 10.1017/S0007114520000252. Epub 2020 Jan 22. PMID 31964428
- [Background] Kolasa, K. M. (1993). The potato and human nutrition. American Potato Journal, 70(5), 375-384. doi:10.1007/BF02849118
- [Background] Liese AD, Nichols M, Sun X, D'Agostino RB Jr, Haffner SM. Adherence to the DASH Diet is inversely associated with incidence of type 2 diabetes: the insulin resistance atherosclerosis study. Diabetes Care. 2009 Aug;32(8):1434-6. doi: 10.2337/dc09-0228. Epub 2009 Jun 1. PMID 19487638
- [Background] Malloy-McFall J, Barkley JE, Gordon KL, Burzminski N, Glickman EL. Effect of the DASH Diet on Pre- and Stage 1 Hypertensive Individuals in a Free-Living Environment. Nutr Metab Insights. 2010 Mar 31;3:15-23. doi: 10.4137/NMI.S3871. eCollection 2010. PMID 23966788
- [Background] Mubarak FM, Froelicher ES, Jaddou HY, Ajlouni KM. Hypertension among 1000 patients with type 2 diabetes attending a national diabetes center in Jordan. Ann Saudi Med. 2008 Sep-Oct;28(5):346-51. doi: 10.5144/0256-4947.2008.346. PMID 18779643
- [Background] Muraki I, Rimm EB, Willett WC, Manson JE, Hu FB, Sun Q. Potato Consumption and Risk of Type 2 Diabetes: Results From Three Prospective Cohort Studies. Diabetes Care. 2016 Mar;39(3):376-84. doi: 10.2337/dc15-0547. Epub 2015 Dec 17. PMID 26681722
- [Background] Nguyen H, Odelola OA, Rangaswami J, Amanullah A. A review of nutritional factors in hypertension management. Int J Hypertens. 2013;2013:698940. doi: 10.1155/2013/698940. Epub 2013 Apr 10. PMID 23691281
- [Background] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Hu EA, Martinez-Gonzalez MA, Salas-Salvado J, Corella D, Ros E, Fito M, Garcia-Rodriguez A, Estruch R, Aros F, Fiol M, Lapetra J, Serra-Majem L, Pinto X, Ruiz-Canela M, Razquin C, Bullo M, Sorli JV, Schroder H, Rebholz CM, Toledo E; PREDIMED Study and SUN Project Investigators. Potato Consumption Does Not Increase Blood Pressure or Incident Hypertension in 2 Cohorts of Spanish Adults. J Nutr. 2017 Dec;147(12):2272-2281. doi: 10.3945/jn.117.252254. Epub 2017 Oct 18. PMID 29046405
- [Background] Svetkey LP, Sacks FM, Obarzanek E, Vollmer WM, Appel LJ, Lin PH, Karanja NM, Harsha DW, Bray GA, Aickin M, Proschan MA, Windhauser MM, Swain JF, McCarron PB, Rhodes DG, Laws RL. The DASH Diet, Sodium Intake and Blood Pressure Trial (DASH-sodium): rationale and design. DASH-Sodium Collaborative Research Group. J Am Diet Assoc. 1999 Aug;99(8 Suppl):S96-104. doi: 10.1016/s0002-8223(99)00423-x. PMID 10450301
- [Background] Venugopal, K., & Mohammed, M. (2014). Prevalence of hypertension in type-2 diabetes mellitus. CHRISMED Journal of Health and Research, 1(4), 223-227. doi:10.4103/2348-3334.142981 38 45 44
- [Background] Vinson JA, Demkosky CA, Navarre DA, Smyda MA. High-antioxidant potatoes: acute in vivo antioxidant source and hypotensive agent in humans after supplementation to hypertensive subjects. J Agric Food Chem. 2012 Jul 11;60(27):6749-54. doi: 10.1021/jf2045262. Epub 2012 Feb 6. PMID 22224463
- [Background] Whelton SP, Hyre AD, Pedersen B, Yi Y, Whelton PK, He J. Effect of dietary fiber intake on blood pressure: a meta-analysis of randomized, controlled clinical trials. J Hypertens. 2005 Mar;23(3):475-81. doi: 10.1097/01.hjh.0000160199.51158.cf. PMID 15716684
- [Background] Zaheer K, Akhtar MH. Potato Production, Usage, and Nutrition--A Review. Crit Rev Food Sci Nutr. 2016;56(5):711-21. doi: 10.1080/10408398.2012.724479. PMID 24925679
- [Background] Zhang Y, You D, Lu N, Duan D, Feng X, Astell-Burt T, Zhu P, Han L, Duan S, Zou Z. Potatoes Consumption and Risk of Type 2 Diabetes: A Meta-analysis. Iran J Public Health. 2018 Nov;47(11):1627-1635. PMID 30581777
- [Background] Zou P, Dennis CL, Lee R, Parry M. Dietary Approach to Stop Hypertension with Sodium Reduction for Chinese Canadians (DASHNa-CC): A Pilot Randomized Controlled Trial. J Nutr Health Aging. 2017;21(10):1225-1232. doi: 10.1007/s12603-016-0861-4. PMID 29188883